CLINICAL TRIAL: NCT00103415
Title: Randomized Clinical Trial Investigating the Effect of Different Exercise Forms on Depression
Brief Title: Trial Investigating the Effect of Different Exercise Forms on Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Demostudiet (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KF01-213/04
Record Dates: First submitted 2005-02-08; First posted 2005-02-09 (Estimated); Last update posted 2006-07-13 (Estimated); Status verified 2005-02

CONDITIONS: Depression
Keywords: Depression; Exercise; Job
MeSH Terms: conditions — Depression; Motor Activity | interventions — Endurance Training; Resistance Training

INTERVENTIONS:
Behavioral: Endurance training
Behavioral: Weight-lifting training

SUMMARY:
During one year, 5-8% of the population will suffer from major depression. Some of the key symptoms are loss of interest in daily activities, loss of energy and sleeping disturbances. The financial consequences of this disease is estimated to be more than 30 million pounds per year in Great Britain and USA alone. There is an increasing interest in the effect exercise has on depression. Smaller studies indicate that exercise is a good treatment for depression. This study will be a large scale randomized trial and will hopefully bring important knowledge on the effects exercise has on depression.

We will compare the effect endurance training, weight-lifting exercise and a control group has on depressive symptoms after 4 months training, twice a week.

DETAILED DESCRIPTION:
Background The incidence of depression is estimated to 3-5%, with a lifetime prevalence of 17% in western societies. The incidence in patient populations affected by chronic and disabling physical illnesses can be as high as 20%. Depressive symptoms as prolonged feeling of sadness, low self esteem and even suicidal tendencies have consequences to not only the patients' social life, but also shows a correlation between the severity of depression and number of work days lost.Depression is associated with increased risk for conditions such as osteoporoses, cardiovascular diseases and dementia. The global burden of disease reported by WHO and others stated that unipolar depressive disorders was the fourth leading cause of disease burden in terms of lost years of healthy life, and that major depression accounted for 12% of all total years lived with disability in 2000. The economic burden of depression on the national economy in the US was in 2000 estimated to 83,1 billion dollars (31% were direct medical costs, 7% were suicide-related mortality costs and 62% were workplace costs).

In 2001 a meta-analysis of randomized controlled trials comparing exercise with other established treatments for patients diagnosed with depression concluded:" The effectiveness of exercise in reducing symptoms of depression cannot be determined because of a lack of good quality research on clinical populations with adequate follow up". The authors found that the majority of studies did not have blinded outcome assessment, nor were they based on the intent-to-treat principle and most had a short follow-up. In conclusion a summary of the latest reviews on the subject, states that it is likely that exercise has an effect in patients diagnosed with depression, but many of the conducted studies have significant methodological problems, which might have a substantial effect on trial results.Despite the above criticism there have been published trials suggesting that exercise has a positive effect in patients diagnosed with depression. A RCT (n=156, age >50, Hamilton rating scale for depression (HAMD)-17mean= 18,5) from 1999 compares an aerobic exercise program, standard medical treatment (SSRI) and a group receiving both. No significant difference was observed between the groups after 16 weeks of intervention.

A study from 2004 showed an effect of aerobic exercise on depression in light to moderately depressed patients (n=82) not receiving medication. The study compared an exercise program of 17,5 kcal/kg/week (jogging one mile approximately equals 100 kcal) with exercise program of 7,5 kcal/kg/week with a control group. After 12 weeks of intervention the group receiving the most strenuous (17,5 kcal/kg/week) program showed a significant reduction in symptoms compared to the group only doing aerobic exercise similar to 7,5 kcal/kg/week and the control group. No significant difference was observed between the low energy expenditure program and the control group. A recently published study in elderly doing progressive resistance training supports these findings on intensity related effect of exercise on depression.The effect of exercise on endorphin, monoamine levels and neutrophin have been proposed as biological mediators of exercise on depression, as well as psychosocial mechanisms such as an increase of physical self-worth and distraction.

Only one previous study have compared aerobic and non-aerobic exercise forms, which theoretically could be working by different biological mechanisms, such as enhanced serotonergic activity due to enhanced free tryptophan levels in aerobic exercise. This study gives us an opportunity to compare the aerobic with non-aerobic exercise in comparable populations.

Studies like this rarely includes measures of biological parameters. Disturbances in the hypothalamic-pituitary axis with high cortisol levels and the lacking ability to suppress endogen cortisol in response to dexamethasone has long been known to accompany depression. Increased fitness has in experimental models shown to decrease cortisol response to psychological and physical stress. Furthermore, serum prolactin has been used as an indicator of central serotonergic activity which has shown an abnormal response to physical activity in depressed patients.

New evidence for the biological effect of exercise includes the increase of BDNF, which is thought to mediate the positive effect of exercise on cognition in response to physical activity in rodents. The deficits in cognitive function in depressed patients is widely recognized, and cognition has previously been shown to relate to fitness levels in older adults in long term physical intervention. The effect of long term physical intervention on cognitive skills, have to our knowledge never been examined in clinically depressed patients.

On this background we argue that a randomized study based on the intent-to-treat principle, including clinical populations and with a long follow-up is needed to evaluate the efficacy of exercise in patients diagnosed with light to moderate depression, regarding depressive symptoms and lost days from work.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-55
* ICD-10 diagnoses F32.0, F32.1, F33.0, F33.1
* Speak fluent danish

Exclusion Criteria:

* Not able to do exercise
* Drug/alcohol addict
* The patient already engages in more than one hour of weekly exercise.
* The patient has not been working the last 24 months due to depression.
* Suicidal behavior.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300
Dates: Start 2005-02; Study Completion 2007-02

PRIMARY OUTCOMES:
HAMD-17

SECONDARY OUTCOMES:
Remission (<8 HAMD-17)
Response (50% reduction of score on HAMD-17)
Job situation

CONTACTS AND LOCATIONS:
Overall Officials: Merete Nordentoft, M.D, Ph.D., Principal Investigator — Bispebjerg Hospital
Locations (1):
- Psychiatric department, Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Krogh J, Saltin B, Gluud C, Nordentoft M. The DEMO trial: a randomized, parallel-group, observer-blinded clinical trial of strength versus aerobic versus relaxation training for patients with mild to moderate depression. J Clin Psychiatry. 2009 Jun;70(6):790-800. doi: 10.4088/jcp.08m04241. PMID 19573478